CLINICAL TRIAL: NCT05842148
Title: IRONY: lIfe afteR ONcoplastic surgerY
Brief Title: Quality of Life After Conservative Oncoplastic Surgery in Breast Cancer Patients (IRONY: lIfe afteR ONcoplastic surgerY)
Acronym: IRONY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Paolo Orsaria, MD. PhD;, Oncoplastic Breast Surgery Consultant, Campus Bio-Medico University
Other Study IDs: PAR 13.23 OSS
Record Dates: First submitted 2023-04-08; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Oncoplastic Breast Surgery; Therapeutic Mammoplasty; Chest Wall Perforated Flaps; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing oncoplastic surgery with type 1 (unilateral) techniques.: All patients with clinical-instrumental diagnosis of breast cancer, candidates for conservative oncoplastic surgery who give informed consent to the study, will be included in the study.
  Type 1 procedures generally involve a unilateral approach, able to guarantee good resective quality, without a significant alteration of the volume with respect to the contralateral breast.
  Post-surgical histopathological data and any associated postsurgical complications will be collected through the compilation of a database.
  Aesthetic and functional post-surgical results related to the quality of life, as data perceived by the surgeon and by the patient, will be collected through the administration of a questionnaire.
  Interventions: Other: Study and recording of post-surgical clinical and pathological data of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery.; Other: Study and recording of any associated post-surgical complications (of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery.; Other: Study and recording of aesthetic and functional post-surgical results related to the quality of life, as data perceived by the surgeon (technical analysis), and by the patient.
- Patients undergoing oncoplastic surgery with type 2 (bilateral) techniques.: All patients with clinical-instrumental diagnosis of breast cancer, candidates for conservative oncoplastic surgery who give informed consent to the study, will be included in the study.
  Type 2 procedures (therapeutic mammoplasty), offer a greater resective potential, but generally require the use of contralateral surgery to obtain symmetry, simultaneous or delayed.
  Post-surgical histopathological data and any associated postsurgical complications will be collected through the compilation of a database.
  Aesthetic and functional post-surgical results related to the quality of life, as data perceived by the surgeon and by the patient, will be collected through the administration of a questionnaire.
  Interventions: Other: Study and recording of post-surgical clinical and pathological data of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery.; Other: Study and recording of any associated post-surgical complications (of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery.; Other: Study and recording of aesthetic and functional post-surgical results related to the quality of life, as data perceived by the surgeon (technical analysis), and by the patient.

INTERVENTIONS:
Other: Study and recording of post-surgical clinical and pathological data of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery. — Control and review of pathological parameters (oncological radicality resection volume, locoregional extension / TNM / multifocality and tumor biological profile).
Other: Study and recording of any associated post-surgical complications (of patients diagnosed with breast cancer undergoing unilateral or bilateral conservative oncoplastic surgery. — Control and review of post-surgical complications (dehiscence, liponecrosis, infection, seroma, hematoma, fibrosis, scar hypertrophy).
Other: Study and recording of aesthetic and functional post-surgical results related to the quality of life, as data perceived by the surgeon (technical analysis), and by the patient. — Control and review of technical analysis by the surgeon, and of psychosocial well-being, physical discomfort, adverse effects of radiotherapy by the patient collected through the administration of a questionnaire.

SUMMARY:
Evaluation of quality of life after conservative oncoplastic surgery in patients with breast cancer

DETAILED DESCRIPTION:
The aim of the study is the evaluation of the oncological, aesthetic and functional results after conservative oncoplastic breast surgery using unilateral or bilateral remodeling techniques in a prospective sample of 250 patients.

Endpoints:

* evaluation of post-surgical histopathological data with a selective focus on the achievement of oncological radicality in relation to the surgical technique ( resection volume, locoregional extension / TNM / multifocality and tumor biological profile) and any major , minor, delayed associated complications (dehiscence, liponecrosis, infection, seroma, hematoma, fibrosis, scar hypertrophy).This data will be collected through the compilation of a database by the health personnel.
* evaluation of aesthetic and functional results related to the quality of life after oncoplastic conservative surgery (unilateral or bilateral), as data perceived by the surgeon (technical analysis), and by the patient (psychosocial well-being, physical discomfort, adverse effects of radiotherapy). This data will be collected through the administration of a questionnaire whose data will be entered into the database by the healthcare personnel.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer
* Must be able for conservative oncoplastic surgery with type 1 and 2 procedures who give informed consent to the study.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients in emergency situations
* Subjects unable to understand and want

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with clinical-instrumental diagnosis of breast cancer, candidates for conservative oncoplastic surgery with type 1 and 2 procedures who give informed consent to the study, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of post-surgical data | three years
  focus on the achievement of oncological radicality in relation to the surgical technique (yes or no).
evaluation of resection volumes | three years
  focus on the resection volume in relation to the surgical technique (cm3).
evaluation of post-surgical staging criteria | three years
  focus on the locoregional extension (TNM staging criteria, American Joint Committee on Cancer, 8th edition)
evaluation of multifocality | three years
  focus on the multifocality (yes or no).
evaluation of tumor biological profile | three years
  focus on the tumor biological profile ( luminal A, luminal B HER2-, luminal B HER2+, HER2+, triple-negative).
evaluation of any post-surgical associated complications | three years
  focus on any major , minor, delayed associated complications (dehiscence, liponecrosis, infection, seroma, hematoma, fibrosis, scar hypertrophy).

SECONDARY OUTCOMES:
evaluation of post-surgical aesthetic results | three years
  focus on data perceived by the surgeon (technical analysis) through a questionnaire with scores ranging from 1 to 3.
evaluation of post-surgical functional results related to the quality of life after oncoplastic conservative surgery (unilateral or bilateral) through a questionnaire with scores ranging from 1 to 3. | three years
  focus on data perceived by the patient (psychosocial well-being, physical discomfort, adverse effects of radiotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Orsaria, Surgeon;, Principal Investigator — Policlinico Universitario Campus Bio-Medico
Locations (1):
- Paolo Orsaria, MD. PhD; [porsaria], Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Orsaria P, Grasso A, Caggiati L, Altomare M, Altomare V. Update on oncoplastic techniques in breast conserving surgery: algorithms for predictable results and custom-made reconstructions. Minerva Surg. 2021 Dec;76(6):512-525. doi: 10.23736/S2724-5691.21.08976-0. Epub 2021 Aug 2. PMID 34338466
- [Background] Cali Cassi L, Vanni G, Petrella G, Orsaria P, Pistolese C, Lo Russo G, Innocenti M, Buonomo O. Comparative study of oncoplastic versus non-oncoplastic breast conserving surgery in a group of 211 breast cancer patients. Eur Rev Med Pharmacol Sci. 2016 Jul;20(14):2950-4. PMID 27460720
- [Background] Orsaria P, Grasso A, Soponaru G, Carnevale F, Scorsone V, Ippolito E, Pantano F, Sammarra M, Piccolo C, Altomare M, Perrone G, Altomare V. Subaxillary Replacement Flap Compared with the Round Block Displacement Technique in Oncoplastic Breast Conserving Surgery: Functional Outcomes of a Feasible One Stage Reconstruction. Curr Oncol. 2022 Nov 30;29(12):9377-9390. doi: 10.3390/curroncol29120736. PMID 36547150
- [Background] Orsaria P, Grasso A, Ippolito E, Pantano F, Sammarra M, Altomare C, Cagli B, Costa F, Perrone G, Soponaru G, Caggiati L, Vanni G, Buonomo OC, Altomare V. Clinical Outcomes Among Major Breast Cancer Subtypes After Neoadjuvant Chemotherapy: Impact on Breast Cancer Recurrence and Survival. Anticancer Res. 2021 May;41(5):2697-2709. doi: 10.21873/anticanres.15051. PMID 33952501